CLINICAL TRIAL: NCT01851239
Title: Venous Thromboembolism Prophylaxis in Medical and Surgical ICUs in a Single University Hospital
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2013-0002
Record Dates: First submitted 2013-04-25; First posted 2013-05-10 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism Prophylaxis; ICU
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- medical ICU inpatients
- surgical ICU inpatients

SUMMARY:
Venous thromboembolism(VTE) is the third most common cardiovascular complication among hospitalized patients, and can even cause death. VTE often occurs in intensive care patients and there had been many efforts to prevent such complication. The American College of Chest Physicians (ACCP) had published evidence-based clinical practice guideline for VTE prophylaxis.

This study focuses on how VTE prophylaxis is being performed in both medical and surgical ICUs in a single University hospital, and sees the differences in such prophylactic patterns.

ELIGIBILITY:
Inclusion Criteria:

* ICU admitted patients

Exclusion Criteria:

* patients under 20 years old

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU admitted patients who are indicated for VTE prophylaxis.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
number of patients prescribed with any measures of VTE prophylaxis in ICU | at the time of ICU admission an expected average of 5 months (When VTE prophylaxis for each patient is being ordered)
  The object of this study is to see the percentage of ICU admitted patients prescribed with VTE prophylaxis, and analyze the adequacy of such prophylactic measure according to the international guideline. Moreover, difference between the VTE prophylaxis pattern of medical and surgical ICUs will also be seek for further analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea